CLINICAL TRIAL: NCT03617354
Title: A Stepped Wedge Cluster Trial to Implement and Evaluate a Model for Training Practising Gynaecologists in Total Laparoscopic Hysterectomy
Brief Title: The Implementation of MinimAlly Invasive Hysterectomy Trial
Acronym: IMAGINE
Status: Completed | Type: Observational
Sponsor: Queensland Centre for Gynaecological Cancer (Other Government)
Responsible Party: Sponsor
Other Study IDs: IMAGINE
Record Dates: First submitted 2018-07-24; First posted 2018-08-06 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Female Reproductive Problem

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Trainee Gynaecologists: 1. RANZCOG accredited O&G specialists who are proficient in RANZCOG laparoscopic skills level 3 or higher;
  2. Surgical capabilities will be assessed using The Global Operative Assessment of Laparoscopic Skills (GOALS) Tool which is an adapted GOALS tool for hysterectomy. GOALS measures depth perception, bimanual dexterity, efficiency, tissue handling and surgeon autonomy each on a 5 point Likert scale. An experienced mentor will assess each surgeon using this scale and skills will be validated against objective outcomes (surgical adverse events recorded in the baseline period).
  3. Will be able to attend each of the 10 training days.
  Interventions: Procedure: Total Laparoscopic Hysterectomy

INTERVENTIONS:
Procedure: Total Laparoscopic Hysterectomy — The trainee gynaecologists are undertaking a training program in performing Total Laparoscopic Hysterectomy

SUMMARY:
Removal of the uterus (hysterectomy) is the most commonly performed major gynaecological procedure in women. Obstetricians and gynaecologist (O&G) surgeons conduct the majority of hysterectomies. Surgical approaches to removal of the uterus include laparoscopic hysterectomy, vaginal hysterectomy with or without laparoscopic assistance and open hysterectomy through an abdominal incision. It is widely accepted that laparoscopic hysterectomy and vaginal hysterectomy are less invasive procedures, cause fewer surgical complications, less postoperative pain, require a shorter hospital stay and are associated with quicker recovery than abdominal hysterectomy. In Australia and despite the evidence, Total Abdominal Hysterectomy (TAH) rates are unreasonably high (~40%) and only 13% of all hysterectomies are done via Total Laparoscopic Hysterectomy (TLH) in Australia.

This study aims to implement and evaluate a training program in TLH for gynaecologists. The potential benefits to the community are:

* A reduction in the incidence of overall surgical adverse events in patients receiving a hysterectomy
* A reduction in the length of hospital stay for patients requiring a hysterectomy
* A reduction in the direct hospital costs for hysterectomy

ELIGIBILITY:
Surgical training program participants Inclusion criteria

1. RANZCOG accredited O&G specialists who are proficient in RANZCOG laparoscopic skills level 3 or higher;
2. Surgical capabilities will be assessed using The Global Operative Assessment of Laparoscopic Skills (GOALS) Tool which is an adapted GOALS tool for hysterectomy. GOALS measures depth perception, bimanual dexterity, efficiency, tissue handling and surgeon autonomy each on a 5 point Likert scale. An experienced mentor will assess each surgeon using this scale and skills will be validated against objective outcomes (surgical adverse events recorded in the baseline period).
3. Will be able to attend each of the 10 training days.

   -

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Trainee gynaecologists
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-03-29 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in proportion of hysterectomy | 36 months
  proportion of hysterectomies performed abdominally through TAH comparing pre-intervention baseline and post-intervention rates

SECONDARY OUTCOMES:
Adverse Events | 36 months
  conversion from TLH to TAH, any anaesthetic incident, intraoperative visceral injury, red cell transfusions, hospital stay greater than 7 days, incidental finding of a malignancy, unplanned readmission, ICU admission or return to theatre, postoperative PE or DVT, development of a fistula, vault haematoma, vaginal vault dehiscence or pelvic infection
Length of hospital stays | 36 months
  days
Cost effectiveness | 36 months
  Cost effectiveness via assessment of: theatre staffing costs; equipment and consumables; Medicare Benefits Schedule items for surgical and anaesthetics fees; costs of health services used after surgery; costs of bed-days; and costs due to readmissions or visits to the emergency department.
Trainee Surgeon proficiency with Total Laparoscopic Hysterectomy | 36 months
  Proficiency is assessed using the Laparoscopic Competency Assessment Tool (L-CAT)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Obermair, Study Chair — Queensland Centre for Gynaecological Cancer
Locations (4):
- Australia (4):
  - Redcliffe Hospital, Brisbane, Queensland
  - Cairns Hospital, Cairns, Queensland
  - Ipswich Hospital, Ipswich, Queensland
  - Mackay Base Hospital, Mackay, Queensland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Obermair A, Armfield NR, Graves N, Gebski V, Hanna GB, Coleman MG, Hughes A, Janda M. How to train practising gynaecologists in total laparoscopic hysterectomy: protocol for the stepped-wedge IMAGINE trial. BMJ Open. 2019 May 9;9(5):e027155. doi: 10.1136/bmjopen-2018-027155. PMID 31072858